CLINICAL TRIAL: NCT01385995
Title: A Controlled Trial of Continuous Positive Airway Pressure (CPAP) Therapy on Metabolic Control in Individuals With Impaired Glucose Tolerance and Sleep Apnea
Brief Title: Effects of Treatment of Sleep Apnea on Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH); Beth Israel Deaconess Medical Center (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Susan Redline, MD, MPH, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HL075077; UL1RR024989 (NIH)
Record Dates: First submitted 2011-06-23; First posted 2011-06-30 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Impaired Glucose Tolerance; Obstructive Sleep Apnea
MeSH Terms: conditions — Glucose Intolerance; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure (CPAP) (Active Comparator)
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) (Philips-Respironics RemStar Pro® CPAP)
- Sham-Continuous Positive Airway Pressure (CPAP) (Sham Comparator)
  Interventions: Device: Sham-Continuous Positive Airway Pressure (CPAP) (Philips-Respironics)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) (Philips-Respironics RemStar Pro® CPAP) — Subjects will be randomized to 8 weeks of CPAP or sham-CPAP, followed by the alternate therapy after a one month wash-out.
  Other Names: Philips-Respironics RemStar Pro® CPAP
  Arms: Continuous Positive Airway Pressure (CPAP)
Device: Sham-Continuous Positive Airway Pressure (CPAP) (Philips-Respironics) — Subjects will be randomized to 8 weeks of CPAP or sham-CPAP, followed by the alternate therapy after a one month wash-out.
  Other Names: Philips-Respironics Sham CPAP
  Arms: Sham-Continuous Positive Airway Pressure (CPAP)

SUMMARY:
The investigators performed a randomized, cross-over controlled clinical trial comparing 8 weeks of Continuous Positive Airway Pressure (CPAP) to 8 weeks of sham-CPAP in patients with moderate to severe Sleep Disordered Breathing (SDB) and impaired glucose tolerance. A rigorous assessment of metabolic responses to SDB treatment in this group is of great clinical significance because this sample is at high risk for developing diabetes. The paradigm shift of CPAP as a mode of prevention can affect clinical practice in the fields of both primary care and sleep medicine.

DETAILED DESCRIPTION:
There are few controlled studies that address whether treatment of sleep apnea improves glucose tolerance. This is a randomized, double-blind cross-over study of subjects with sleep apnea (apnea hypopnea index > 15) and impaired glucose tolerance. Subjects will be randomized to 8 weeks of Continuous Positive Airway Pressure (CPAP) or sham-CPAP, followed by the alternate therapy after a one month wash-out. After each treatment, subjects will undergo 2-hour oral glucose tolerance testing, polysomnography, actigraphy, and measurements of indices of glucose control. The investigators intend to analyze the changes in glucose metabolism and insulin sensitivity in patients with sleep apnea with CPAP intervention.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe Sleep Disordered Breathing (SDB) defined by an Apnea Hypopnea Index (AHI) > 15
* had evidence of Impaired Glucose Tolerance (IGT) defined by the mean 2-hour Oral Glucose Tolerance Test (OGTT) glucose of > 140 mg/dl calculated from the two 2-hour OGTTs performed within 3 days of each other

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, M.D., M.P.H., Study Director — Brigham and Women's Hospital; Faramarz Beigi, Principal Investigator — Case Western Reserve University; H Lester Kirchner, PhD, Principal Investigator — Case Western Reserve University; Carol Rosen, M.D., Principal Investigator — Case Western Reserve University; John Haaga, M.D., Principal Investigator — Case Western Reserve University; Kingman Strohl, M.D., Principal Investigator — Case Western Reserve University; Reena Mehra, M.S., M.S., Principal Investigator — Case Western Reserve University; Denise Babineau, PhD, Principal Investigator — Case Western Reserve University; Tanya Weinstock, M.D., Principal Investigator — Brigham and Women's Hospital

REFERENCES:
- [Derived] Weinstock TG, Wang X, Rueschman M, Ismail-Beigi F, Aylor J, Babineau DC, Mehra R, Redline S. A controlled trial of CPAP therapy on metabolic control in individuals with impaired glucose tolerance and sleep apnea. Sleep. 2012 May 1;35(5):617-625B. doi: 10.5665/sleep.1816. PMID 22547887

RESULTS

PARTICIPANT FLOW:
Period: Period 1, 2 Months
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Sham-Continuous Positive Airway Pressure
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Washout Period, 1 Month
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Sham-Continuous Positive Airway Pressure
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0
Period: Period 2, 2 Months
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Sham-Continuous Positive Airway Pressure
Started | 24 | 25
Completed | 24 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Sham-Continuous Positive Airway Pressure | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 53 (8) | 53.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Normalization of Impaired Glucose Tolerance (IGT)
Description: Number of subjects who experienced normalization of the mean 2-hour oral glucose tolerance test (OGTT) in the overall sample undergoing therapeutic CPAP vs. sham CPAP. (2-hour OGTT glucose< 140 mg/dL)
Time Frame: 20 weeks
Population: All available oral glucose tolerance test data was analyzed for the total sample.
Measure: Number; unit: subjects
Groups:
- Therapeutic CPAP: Assessment of number of subjects with normalization of oral glucose tolerance test from baseline after therapeutic CPAP therapy, in total sample, with the active periods of both sequences combined.
- Sham CPAP: Assessment of number of subjects with normalization of oral glucose tolerance test from baseline after sham CPAP therapy, in total sample, with the sham periods of both sequences combined.
Arm/Group | Therapeutic CPAP | Sham CPAP
Number analyzed (Participants) | 47 | 47
subjects | 7 | 5
Statistical Analysis 1: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent to treat approach a Generalized Estimating Equation (GEE) was used to estimate the effect of therapy (CPAP or Sham) on the odds of normalization of Impaired Glucose Tolerance (IGT). This model provides an estimate of the odds ratio of normalizing the 2-hour oral glucose tolerance test (OGTT) with CPAP compared with Sham-CPAP; Test type: Superiority or Other; p = 0.57, Generalized Estimating Equation; Controlled for period and baseline 2 hour OGTT glucose level; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.52 to 3.24]

2. Secondary Outcome: Mean and Standard Deviation of Glucose Indices After Therapeutic CPAP vs. Sham
Description: Reported values include: fasting glucose (mg/dL), 2 hour Oral Glucose Tolerance Test (OGTT) (mg/dL)
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Therapeutic CPAP | Sham CPAP
Number analyzed (Participants) | 50 | 49
mg/dL
  Fasting Glucose (mg/dL), CPAP | 106.4 (12.4) [-1.2 to 3.0] | 105.6 (13.3)
  2-Hour OGTT (mg/dL), CPAP | 171.1 (43.5) [-16.3 to 1.7] | 178.2 (48.5)
Statistical Analysis 1: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of glucose indices, in this case fasting glucose, between CPAP and sham-CPAP; Test type: Superiority or Other; p = 0.38, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, Apnea-Hypopnea Index (AHI), gender and race; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-1.2 to 3.0]
Statistical Analysis 2: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between measures of glucose indices, in this case, 2 hour OGTT, and therapeutic CPAP vs. Sham; Test type: Superiority or Other; p = 0.11, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-16.3 to 1.7]
Statistical Analysis 3: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of glucose indices, in this case fasting glucose, between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N=25; Test type: Superiority or Other; p = 0.86, Regression, Linear; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.3 to 2.7]
Statistical Analysis 4: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of glucose indices, in this case 2-hour oral glucose tolerance test (OGTT) glucose, between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N= 25; Test type: Superiority or Other; p = 0.08, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = -11.6, 95% CI 2-sided [-24.6 to 1.3]

3. Secondary Outcome: Mean and Standard Deviation of Insulin Indices After Therapeutic CPAP vs. Sham
Description: The data for fasting and 2 hour Insulin (iIU/dL) are presented according to therapeutic CPAP vs. Sham CPAP.
Time Frame: 20 weeks
Population: All subjects with available fasting and and 2-hour insulin measurements are included.
Measure: Mean (Standard Deviation); unit: iIU/dL
Arm/Group | Therapeutic CPAP | Sham CPAP
Number analyzed (Participants) | 50 | 46
iIU/dL
  Fasting Insulin (iIU/dL) | 16.4 (9.0) [-3.4 to 0.5] | 17.2 (10.1)
  2-Hour OGTT Insulin (iU/dL) | 110.1 (60.7) [-23.3 to 2.8] | 114.3 (68.1)
Statistical Analysis 1: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of insulin indices, in this case, fasting insulin, between CPAP and sham-CPAP; Test type: Superiority or Other; p = 0.14, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, Apnea-Hypopnea Index (AHI), gender and race; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.4 to 0.5]
Statistical Analysis 2: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of insulin indices, in this case, 2-hour oral glucose tolerance test (OGTT) insulin, between CPAP and sham-CPAP; Test type: Superiority or Other; p = 0.12, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, Apnea-Hypopnea Index (AHI), gender and race; Mean Difference (Final Values) = -10.7, 95% CI 2-sided [-23.3 to 2.8]
Statistical Analysis 3: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of insulin indices, in this case fasting insulin, between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N=23; Test type: Superiority or Other; p = 0.10, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-5.2 to 0.5]
Statistical Analysis 4: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of insulin indices, in this case oral glucose tolerance test (OGTT) insulin, between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N=23; Test type: Superiority or Other; p = 0.002, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = -28.7, 95% CI 2-sided [-46.5 to -10.9]

4. Secondary Outcome: Mean and Standard Deviation of Indices of Insulin Resistance With Therapeutic CPAP vs. Sham
Description: Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) with therapeutic CPAP vs. Sham CPAP
Time Frame: 20 weeks
Population: All subjects with available fasting insulin, glucose measurements
Measure: Mean (Standard Deviation); unit: percentage of beta cell function
Arm/Group | Therapeutic CPAP | Sham CPAP
Number analyzed (Participants) | 50 | 46
percentage of beta cell function | 4.4 (2.6) [-17.6 to 1.8] | 4.6 (3.0)
Statistical Analysis 1: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and Homeostasis Model Assessment-Insulin Resistance (HOMA-IR), between CPAP and sham-CPAP; Test type: Superiority or Other; p = 0.18, Regression, Linear; Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-17.6 to 3.8]
Statistical Analysis 2: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and measures of insulin resistance, in this case Homeostasis Model Assessment-Insulin Resistance (HOMA-IR), between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N=23; Test type: Superiority or Other; p = 0.08, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = -14.1, 95% CI 2-sided [-27.5 to 1.8]

5. Secondary Outcome: Mean and Standard Deviation of Insulin Sensitivity Index (ISI(0,120)) With Therapeutic CPAP vs. Sham
Description: Insulin Sensitivity Index derived from the Gutt Index, uses the plasma glucose and insulin concentration from fasting (0 min) and 120-min samples from the OGTT, to calculate (Metabolic Clearance Rate)/log (Mean Serum Insulin). The range of possible values is based on the subset ranges of fasting and oral glucose tolerance test (OGTT) insulin and fasting and OGTT glucose, which calculate to be a range of 1.6 to 206.8. An increase in the ISI (0,120) indicates an improvement in the insulin sensitivity.
Time Frame: 20 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapeutic CPAP | Sham CPAP
Number analyzed (Participants) | 49 | 46
units on a scale | 12 (3.3) | 12 (3.8)
Statistical Analysis 1: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and the Insulin Sensivity Index, between CPAP and sham-CPAP; Test type: Superiority or Other; p = 0.20, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, Apnea-Hypopnea Index (AHI), gender and race; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-2.0 to 9.8]
Statistical Analysis 2: Comparison: Therapeutic CPAP vs Sham CPAP; Based on an intent-to-treat approach, a linear mixed effect model was used to estimate the association between therapy and the Insulin Sensitivity Index (ISI(0,120)), between CPAP and sham-CPAP, stratified for the most severe sleep apnea group (Apnea-Hypopnea Index (AHI) >=30) in order to assess whether the differences in the effect of CPAP on outcomes were observed according to sleep apnea severity. N=23; Test type: Superiority or Other; p = 0.002, Regression, Linear; Adjusted for period, baseline level of the outcome variable, BMI, AHI, gender and race; Mean Difference (Final Values) = 13.3, 95% CI 2-sided [5.2 to 22.1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Continuous Positive Airway Pressure (CPAP) | Sham-Continuous Positive Airway Pressure
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50
Other Adverse Events (participants affected / at risk) | 12/50 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Positive Airway Pressure (CPAP) (N=50) | Sham-Continuous Positive Airway Pressure (N=50)
Chest Pain (non cardiac) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Positive Airway Pressure (CPAP) (N=50) | Sham-Continuous Positive Airway Pressure (N=50)
skin irritation from nasal CPAP mask (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Boil on Lip (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Drowsy Driving (Social circumstances) | 0 (0) | 1 (1) — Deemed to be unrelated to study; direct result from sleep deprivation; event last less than 5 seconds.
Claustrophobia (Psychiatric disorders) | 0 (0) | 1 (1) — secondary to mask
Skin irritation from echocardiogram leads (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) — While wearing mask

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes